CLINICAL TRIAL: NCT00536354
Title: Effects Of Postural Orientation In The Use Of School Backpacks In Elementary School Students
Brief Title: Postural Orientation In The Use Of School Backpacks
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SFernandes
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Backpain; Prevention; Physical Therapy
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Postural Orientation

SUMMARY:
This study will examine the effects of postural orientation in the use of school backpacks among elementary school students.

ELIGIBILITY:
Inclusion Criteria:

* Children from seven to ten years of age. Studing in private elementary school.

Ages: 7 Years to 10 Years | Sex: All
Age Groups: Child
Dates: Start 2005-08; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susi MS Fernandes, Master, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil